CLINICAL TRIAL: NCT00561418
Title: Histone Deacetylase (HDAC) Inhibition Using Vorinostat (SAHA) After Autologous Hematopoietic Stem Cell Transplantation for High Risk Lymphoma
Brief Title: Vorinostat After Stem Cell Transplant in Treating Patients With High-Risk Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Craig Hofmeister, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07047; NCI-2011-03145 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Lymphoma; Small Intestine Cancer
Keywords: recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult Hodgkin lymphoma; recurrent mantle cell lymphoma; adult nasal type extranodal NK/T-cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; small intestine lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Hodgkin Disease; Lymphoma, Mantle-Cell; Lymphoma, Extranodal NK-T-Cell; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat (SAHA) (Experimental): Vorinostat (SAHA) will be administered orally starting approximately day +60 post HSCT for 21 consecutive days of a 28-day cycle for up to a maximum of 11 cycles with the dose escalations.
  Interventions: Drug: vorinostat; Other: Correlative studies

INTERVENTIONS:
Drug: vorinostat — Vorinostat (SAHA) will be administered orally starting approximately day +60 post HSCT for 21 consecutive days of a 28-day cycle for up to a maximum of 11 cycles.
  Other Names: SAHA
Other: Correlative studies — Laboratory as well as quality of life correlative studies will be obtained at days +26 to +38 (at approximately 1 month post HSCT),days +56 to +66 (≈2 mos), and at Cycle 2 Day 1 (≈3 mos.), Cycle 3 Day 1 (≈4 mos.), Cycle 5 Day 1 (≈6 mos.),Cycle 7 Day 1 (≈8 mos.), and off study (ideally at ≈12 mos.)

SUMMARY:
RATIONALE: Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth, and may stimulate the immune system to stop cancer cells from growing.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat after stem cell transplant in treating patients with high-risk lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess dose-limiting and nonhematologic toxicity of prolonged administration of vorinostat (SAHA) when administered after autologous peripheral blood stem cell transplantation in patients with high-risk lymphoma.

Secondary

* To determine, preliminarily, clinical activity by assessing the overall survival and progression-free survival.
* To evaluate the effect of vorinostat on immune reconstruction and acetylation.
* To obtain pilot data regarding an association of vorinostat with patient quality of life and inflammatory cytokine production of peripheral blood mononuclear cells.

OUTLINE: This is a dose-escalation study of vorinostat (SAHA).

Approximately 60 days after autologous hematopoietic stem cell transplantation (HSCT), patients receive oral vorinostat once daily on days 1-21. Treatment repeats every 28 days for up to 11 courses in the absence of unacceptable toxicity or disease progression.

Blood and bone marrow samples are collected periodically for laboratory correlative studies comprising immune reconstitution assays, regulatory T-cell expansion analysis, H3 and H4 acetylation by immunohistochemistry, cytokine bead array to quantify interleukin (IL)-2, IL-4, IL-5, IL-6, IL-10, tumor necrosis factor alpha and interferon gamma. Quality of life correlative studies are measured by questionnaires periodically.

After completion of study treatment, patients are followed for at least 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have received a BEAM (cytarabine, etoposide, melphalan, carmustine)-conditioned autologous stem cell transplantation for any of the following high-risk lymphomas:

  * Diffuse large B-cell lymphoma as defined by:

    * Induction failure but with response to salvage therapy
    * Relapse less than one year after completion of induction therapy
    * Elevated lactate dehydrogenase (LDH) at relapse
    * Stage III/IV disease at relapse
    * Positive PET scan after induction or salvage therapy
    * Age ≤ 75 and ≥ 60 years
  * Follicular lymphoma as defined by:

    * Progressive disease after two or more prior regimens
    * Transformed to aggressive lymphoma but still chemotherapy sensitive
    * Not felt to be a good candidate for an allogeneic transplantation
  * Hodgkin lymphoma as defined by:

    * Primary refractory disease
    * Relapse less than one year after completion of induction therapy
    * Relapse with PET-positive disease after salvage therapy
    * Relapsed refractory and not felt to be a good candidate for an allogeneic transplantation
  * Mantle cell lymphoma

    * Chemotherapy-sensitive disease after induction therapy
    * Chemotherapy-sensitive relapsed disease and not felt to be a good candidate for an allogeneic transplantation
  * T-cell non-Hodgkin lymphoma (NHL)

    * Peripheral T-cell lymphoma not otherwise specified and one or more of the following at diagnosis:

      * High LDH
      * Marrow involvement
      * Age > 60 years
      * Low platelet count
      * Relapsed chemotherapy-sensitive disease
    * Angioimmunoblastic lymphadenopathy with dysproteinemia
    * Anaplastic lymphoma kinase-negative anaplastic NHL
    * Enteropathy-associated T-cell NHL
    * Natural killer (NK)/T-cell NHL and stage III/IV disease at diagnosis
    * NK blastic NHL

PATIENT CHARACTERISTICS:

* ECOG (Eastern Cooperative Oncology Group) /WHO performance status 0-2
* ANC (absolute neutrophil count) ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 1.5 mg/dL
* AST (aspartate aminotransferase)/ALT (Alanine transaminase) ≤ 2 x upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 50 mL/min
* No severe or uncontrolled systemic illness
* Patients must be able to swallow capsules
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use at least two adequate barrier methods of contraception during study and for 90 days after completion of study therapy
* No other malignancy within the past 5 years other than nonmelanoma skin cancer, carcinoma in situ of the cervix, or a malignancy considered by their physician to be at less than 30% risk of relapse
* No congenital long QT syndrome
* No significant history of uncontrolled cardiac disease (i.e., uncontrolled hypertension, unstable angina, myocardial infarction within the past 6 months, or uncontrolled congestive heart failure)
* No active bacterial, fungal, or viral infection
* No known HIV infection
* No active hepatitis B and/or hepatitis C infection
* No other medical condition, including mental illness or substance abuse, deemed by the Investigator(s) to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

PRIOR CONCURRENT THERAPY:

* Recovered from the majority of the toxicities from the autologous transplantation (must have returned to their pretransplant baseline or have no greater than grade I extramedullary toxicity Common Toxicity Criteria for Adverse Effects[CTCAE 3.0])
* No prior treatment with a histone deacetylase (HDAC) inhibitor (e.g., depsipeptide, MS-275, LAQ-824, belinostat, valproic acid)
* More than 4 weeks since prior and no concurrent class Ia, Ib, or Ic antiarrhythmic drugs
* No other concurrent antineoplastic chemotherapy or biologic therapy
* No concurrent radiotherapy, unless for local control of bone pain

  * Irradiated area for pain management should be as small as possible and lesions within the irradiated field cannot be used for response
* No concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and antitumor activity of vorinostat (SAHA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig C. Hofmeister, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Hofmeister CC, Williams N, Geyer S, Hade EM, Bowers MA, Earl CT, Vaughn J, Bingman A, Humphries K, Lozanski G, Baiocchi RA, Jaglowski SM, Blum K, Porcu P, Flynn J, Penza S, Benson DM, Andritsos LA, Devine SM. A phase 1 study of vorinostat maintenance after autologous transplant in high-risk lymphoma. Leuk Lymphoma. 2015 Apr;56(4):1043-9. doi: 10.3109/10428194.2014.963073. Epub 2014 Nov 20. PMID 25213183
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat (SAHA): Vorinostat (SAHA) will be administered orally starting approximately day +60 post HSCT for 21 consecutive days of a 28-day cycle for up to a maximum of 11 cycles with the dose escalations.
  vorinostat: Vorinostat (SAHA) will be administered orally starting approximately day +60 post HSCT for 21 consecutive days of a 28-day cycle for up to a maximum of 11 cycles.
  Correlative studies: Laboratory as well as quality of life correlative studies will be obtained at days +26 to +38 (at approximately 1 month post Hematopoietic Stem Cell Transplantation),days +56 to +66 (≈2 mos), and at Cycle 2 Day 1 (≈3 mos.), Cycle 3 Day 1 (≈4 mos.), Cycle 5 Day 1 (≈6 mos.),Cycle 7 Day 1 (≈8 mos.), and off study (ideally at ≈12 mos.)
Period: Overall Study
Arm/Group | Vorinostat (SAHA)
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat (SAHA): Vorinostat (SAHA) will be administered orally starting approximately day +60 post HSCT for 21 consecutive days of a 28-day cycle for up to a maximum of 11 cycles with the dose escalations.
  vorinostat: Vorinostat (SAHA) will be administered orally starting approximately day +60 post HSCT for 21 consecutive days of a 28-day cycle for up to a maximum of 11 cycles.
  Correlative studies: Laboratory as well as quality of life correlative studies will be obtained at days +26 to +38 (at approximately 1 month post HSCT),days +56 to +66 (≈2 mos), and at C2D1 (≈3 mos.), C3D1 (≈4 mos.), C5D1 (≈6 mos.),C7D1 (≈8 mos.), and off study (ideally at ≈12 mos.)
Arm/Group | Vorinostat (SAHA)
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 55 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Vorinostat (SAHA) After Autologous Stem Cell Transplantation
Description: NCI CTCAE version 3.0 was used to assess Adverse Events (AE) Grade 1=Mild AE Grade 2=Moderate AE Grade 3=Severe AE Grade 4=Life-threatening or disabling AE
Time Frame: Up to 3 years
Measure: Number; unit: patients
Arm/Group | Vorinostat (SAHA)
Number analyzed (Participants) | 23
patients
  Fatigue (Grade 1, 2) | 12
  Lymphopenia (Grade 1-4) | 11
  Thrombocytopenia (Grade 1-3) | 11
  Leukopenia (Grade 1-3) | 10
  Anemia (Grade 1-3) | 10

2. Secondary Outcome: Clinical Benefit
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Population: Response following AHSCT
Measure: Number; unit: patients
Arm/Group | Vorinostat (SAHA)
Number analyzed (Participants) | 23
patients
  Complete Response (CR) | 13
  Partial Response (PR) | 3
  Stable Disease(SD) | 2
  Not evaluable | 5

3. Secondary Outcome: Duration of Response
Description: Median follow up of living patients
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Vorinostat (SAHA)
Number analyzed (Participants) | 18
months | 23.2 [8.7 to 58.8]

4. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 3 years
Population: Unable to calculate time to progression for patients due to not enough follow up time
Arm/Group | Vorinostat (SAHA)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was utilized for adverse event reporting.
Arm/Group | Vorinostat (SAHA)
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 12/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (SAHA) (N=23)
fatigue (Investigations) | 12 (12)
Lymphopenia (Investigations) | 11 (11)
Thrombocytopenia (Injury, poisoning and procedural complications) | 11 (11)
Leukopenia (Investigations) | 10 (10)
anemia (Blood and lymphatic system disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes